CLINICAL TRIAL: NCT06310902
Title: Single-cell Sequencing Analysis of Resectable/Borderline Resectable Pancreatic Cancer Patients
Status: Recruiting | Type: Observational
Sponsor: Fujian Medical University Union Hospital (Other)
Responsible Party: Principal Investigator, Yu Pan, Principal Investigator, Fujian Medical University Union Hospital
Other Study IDs: 2024KY022
Record Dates: First submitted 2024-03-06; First posted 2024-03-15 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Pancreatic Neoplasms
Keywords: Pancreatic neoplasms; Single-cell sequencing; Immune microenvironment
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — tumor tissue, paracancerous tissue, blood, and lymphonodu
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Borderline Resectable Pancreatic Cancer: Cancer tissue specimens can be collected postoperatively following neoadjuvant chemotherapy.
  Interventions: Diagnostic Test: Single-cell Sequencing Analysis
- Resectable Pancreatic Cancer: Cancer tissue specimens can be directly collected postoperatively
  Interventions: Diagnostic Test: Single-cell Sequencing Analysis

INTERVENTIONS:
Diagnostic Test: Single-cell Sequencing Analysis — Identification of rare cell populations, the characterization of cell types and subtypes, and the discovery of novel cell states.

SUMMARY:
Preoperative neoadjuvant chemotherapy is widely used in treating patients with borderline resectable pancreatic cancer (BRPC). However, there are limitations in this field. Treatment strategies and definitions for BRPC patients differ, and the efficacy and prognosis of neoadjuvant chemotherapy vary greatly.This study aims to utilize single-cell sequencing technology to investigate in-depth the composition and interactions of the tumor microenvironment in patients from the surgical-only group and the preoperative neoadjuvant chemotherapy group.

ELIGIBILITY:
Inclusion Criteria:

* 18 years ≤ age ≤ 75 years.
* Resectable/borderline resectable pancreatic cancer patients diagnosed based on pathological and preoperative imaging evaluation.
* No prior history of any form of anti-tumor treatment.
* At least one measurable lesion.
* Eastern Cooperative Oncology Group (ECOG): 0-1.
* Not participated in any other clinical studies before or during treatment.
* Willingness to participate voluntarily in this study, signing an informed consent form.

Exclusion Criteria:

* History of any other malignant tumor, except for completely resected basal cell or squamous cell carcinoma of the skin or carcinoma in situ of the cervix, within the past 5 years.
* Vaccination with live vaccines within 4 weeks prior to enrollment or during the study period.
* Active autoimmune diseases or a history of autoimmune diseases within the past 4 weeks before enrollment.
* Allogeneic bone marrow or organ transplantation.
* Active gastric or duodenal ulcers, ulcerative colitis, or active bleeding from unresected tumors in the gastrointestinal tract, or other conditions determined by the investigator that may cause gastrointestinal bleeding or perforation.
* Evidence or history of significant bleeding tendency within 3 months prior to enrollment (bleeding >30 mL within 3 months, hematemesis, melena, or hematochezia), hemoptysis (>5 mL of fresh blood within 4 weeks), or occurrence of thromboembolic events within 12 months (including stroke events and/or transient ischemic attacks).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Resectable/borderline resectable pancreatic cancer patients diagnosed based on pathological and preoperative imaging evaluation
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Bioinformatics analysis of single-cell sequencing results | Collected during surgical treatment
  Using single-cell sequencing technology, in-depth analysis of surgical samples from resectable/borderline resectable pancreatic cancer patients is conducted to investigate the composition and interactions of the tumor microenvironment in pancreatic cancer.

CONTACTS AND LOCATIONS:
Locations (1):
- Fujian Medical University Union Hospital, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data (IPD) available to other researchers

REFERENCES:
- [Background] Versteijne E, van Dam JL, Suker M, Janssen QP, Groothuis K, Akkermans-Vogelaar JM, Besselink MG, Bonsing BA, Buijsen J, Busch OR, Creemers GM, van Dam RM, Eskens FALM, Festen S, de Groot JWB, Groot Koerkamp B, de Hingh IH, Homs MYV, van Hooft JE, Kerver ED, Luelmo SAC, Neelis KJ, Nuyttens J, Paardekooper GMRM, Patijn GA, van der Sangen MJC, de Vos-Geelen J, Wilmink JW, Zwinderman AH, Punt CJ, van Tienhoven G, van Eijck CHJ; Dutch Pancreatic Cancer Group. Neoadjuvant Chemoradiotherapy Versus Upfront Surgery for Resectable and Borderline Resectable Pancreatic Cancer: Long-Term Results of the Dutch Randomized PREOPANC Trial. J Clin Oncol. 2022 Apr 10;40(11):1220-1230. doi: 10.1200/JCO.21.02233. Epub 2022 Jan 27. PMID 35084987
- [Background] Gonzalez-Silva L, Quevedo L, Varela I. Tumor Functional Heterogeneity Unraveled by scRNA-seq Technologies. Trends Cancer. 2020 Jan;6(1):13-19. doi: 10.1016/j.trecan.2019.11.010. Epub 2020 Jan 3. PMID 31952776
- [Result] Versteijne E, Suker M, Groothuis K, Akkermans-Vogelaar JM, Besselink MG, Bonsing BA, Buijsen J, Busch OR, Creemers GM, van Dam RM, Eskens FALM, Festen S, de Groot JWB, Groot Koerkamp B, de Hingh IH, Homs MYV, van Hooft JE, Kerver ED, Luelmo SAC, Neelis KJ, Nuyttens J, Paardekooper GMRM, Patijn GA, van der Sangen MJC, de Vos-Geelen J, Wilmink JW, Zwinderman AH, Punt CJ, van Eijck CH, van Tienhoven G; Dutch Pancreatic Cancer Group. Preoperative Chemoradiotherapy Versus Immediate Surgery for Resectable and Borderline Resectable Pancreatic Cancer: Results of the Dutch Randomized Phase III PREOPANC Trial. J Clin Oncol. 2020 Jun 1;38(16):1763-1773. doi: 10.1200/JCO.19.02274. Epub 2020 Feb 27. PMID 32105518